CLINICAL TRIAL: NCT05273918
Title: Monitoring and Evaluation of a Cognitive Behavioral Therapy Program Focused on Attention and Emotion Regulation for Children With Fetal Alcohol Spectrum Disorder
Acronym: SEPAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: logistic problem and absence of coordinating Investigator
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/CHU/06
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Fetal Alcohol Spectrum Disorders; Hyperactivity Disorder; Attention Deficit
Keywords: FASD; ADHD
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy cognitivo-comportmental (Experimental): Each child will participate in a structured cognitive behavioral therapy program entitled "better manage your anger and frustration". 15 workshops is planned.
  Interventions: Other: cognitivo-comportmental therapy
- Body mediation (Active Comparator): Each child will participate in sports, artistic or fun activities involving the body (physical, emotional and communicative dimensions)
  Interventions: Other: body mediation

INTERVENTIONS:
Other: cognitivo-comportmental therapy — 15 workshops once a week during 90 minutes
  Arms: Therapy cognitivo-comportmental
Other: body mediation — 15 workshops once a week during 90 minutes
  Arms: Body mediation

SUMMARY:
This is a multi-center, prospective, randomized, open-label, controlled trial with two parallel arms and blinded endpoint assessment.

It aims yo compare the 6-month efficacy of a group CBT program versus body-mediated intervention (meditation) children (7-13 years) with ADHD-associated FASD and emotional dysregulation via a measurement of the Aggressive Behaviors subscale score of the Dysregulation Profile subset of the CBCL scale.

ELIGIBILITY:
Inclusion Criteria:

* child with fetal alcohol spectrum disorder
* child with attention deficit disorder with / without hyperactivity
* child with a score upper than or equal to 180 points on the "Aggressive behavior", "Anxiety / Depression" and "Concentration problems" subscales of the CBCL
* child followed in La Reunion, Montpellier or Bordeaux University Hospital
* child whose parents are affiliated with social security
* child who accepts to participate and whose parents have given their consent

Exclusion Criteria:

* non-french speaking child or parents / non-creole speaking child or parents
* child who already participate to CBT or body mediation groups

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
effectiveness of cognitive behavioral therapy program | 7 months after inclusion
  score on Child Behavior Check List (CBCL) scale. Minimum value = 50 (normal) and maximal value = 100 (pathologic). Score between 50 and 65 is mormal and score between 70 and 100 is pathologic and needs patients medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Michel SPODENKIEWICZ, MD, Principal Investigator — CHU de La Réunion
Locations (3):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - CHU de Montpellier - Hôpital Saint Eloi, Montpellier
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No